CLINICAL TRIAL: NCT00664261
Title: Addressing Parental Smoking by Changing Pediatric Office Systems
Brief Title: Clinical Effort Against Secondhand Smoke (CEASE) Program or Standard Care in Helping Parents Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Health Services Research
Other Study IDs: CDR0000584270; MGH-200P002323
Record Dates: First submitted 2008-04-19; First posted 2008-04-22 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2011-06

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Counseling; Early Intervention, Educational

INTERVENTIONS:
Behavioral: smoking cessation intervention
Other: cancer prevention
Other: counseling intervention
Other: educational intervention
Other: laboratory biomarker analysis
Other: questionnaire administration
Other: survey administration
Procedure: study of high risk factors

SUMMARY:
RATIONALE: The Clinical Effort Against Secondhand Smoke (CEASE) program may be more effective than standard care in increasing the number of parents who stop smoking.

PURPOSE: This randomized clinical trial is studying how well the CEASE program works compared with standard care in helping parents stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the effectiveness of the Clinical Effort Against Secondhand Smoke (CEASE) intervention vs no intervention in increasing clinicians' delivery of evidence-based parental smoking cessation assistance in pediatric healthcare settings.
* To compare the effectiveness of this intervention vs no intervention on parental smoking behaviors.
* To test the level of systematic practice implementation of the intervention using existing validated measures in an Implementation Process Survey (IPS).
* To evaluate, in an exploratory fashion, additional key implementation step measures mapped from the five A's (Ask, Advise, Assess, Assist, Arrange) to see how well they predict tobacco control service delivery in pediatric healthcare settings.
* To use process results from the IPS (i.e., previously validated and exploratory measures) to improve the adoption, implementation, and maintenance of the intervention in this study.

OUTLINE: This is a multicenter study. Participants are stratified according to practice. Participants are randomized to 1 of 2 intervention arms.

* Arm I (Clinical Effort Against Secondhand Smoke [CEASE] intervention): The CEASE intervention incorporates a number of materials into the operations of the pediatric practice, including baseline questionnaires that screen for parental tobacco use and readiness to quit smoking, enroll in quitline counseling, or explore pharmacotherapy; a label that affixes to the child's problem list in the medical record, documenting parental smoking status and indicating the patient's secondhand exposure, thus encouraging continuity of cessation support in cross-coverage situations; and decision support for clinicians that prompts delivery of exposure-reduction counseling and distribution of motivational-messaging handouts (i.e., halflets) to parents for education, skills training, and psychosocial support. Parental messaging elements include strategies or methods for quitting, collaborative goal setting, identifying personal barriers to quitting, and focused strategies for reducing secondhand-smoke exposure of the patient. Additional intervention materials include a HIPAA-compliant form for enrolling the smoker in counseling through the telephone quitline; pre-printed, practice-embossed prescription pads for prescribing over-the-counter nicotine-replacement therapy when desired by the smoker; pharmacotherapy posters in pediatric patient examination rooms to inform parental smokers and assist clinicians in discussing tobacco dependence treatment; and a simple implementation guide to support integrating the parent, clinician, and practice levels of the intervention.

The CEASE intervention also incorporates telephone counseling after the pediatric healthcare visit to ensure that parents receive professional, ongoing smoking-cessation counseling. Parental smokers undergo an exit interview survey and follow-up telephone surveys at 3 months and 12 months for evaluation of content of tobacco control delivered during the visit; use of messaging materials, medications, and telephone counseling sessions; current smoking status; and rules about smoking in the home and car. If the parent has had a 7-day quit at the 12-month follow-up, the parent is also asked to provide a saliva sample for cotinine analysis to confirm nonsmoking status.

* Arm II (control): Participants complete a questionnaire at baseline and an exit interview survey. They also complete telephone interviews at 3 month and 12 months. If the parent has had a 7-day quit at the 12-month follow-up, the parent is also asked to provide a saliva sample for cotinine analysis to confirm nonsmoking status.

In both arms, participating practitioners and key office staff complete Implementation Process Surveys at baseline and at 6 weeks and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Parents or guardians meeting the following criteria:

  * Self-identified as smokers on the baseline survey
  * Must have a child who is seen by a pediatrician in a participating practice

    * Child must not have a medically emergent condition that requires transfer outside the practice for immediate medical intervention
  * Must be present at the child's healthcare visit
* Pediatric practice meeting the following criteria:

  * Participates in the Pediatric Research in Office Settings (PROS) network
  * Practice manager and a majority of pediatricians are willing to implement a tobacco control strategy for parental smokers
  * Cares for at least 2,000 families
  * Located in a geographically distinct location to minimize contamination effects of the intervention

    * No practices at the same geographic location

PATIENT CHARACTERISTICS:

* Have a telephone at home (parent or guardian)
* Able to speak English (parent or guardian)
* Have a working fax machine (practice)

PRIOR CONCURRENT THERAPY:

* No prior enrollment in this study during a previous visit to the pediatric healthcare clinician (parent or guardian)
* No prior participation in phase II focus groups or other pilot tobacco control studies (practice)
* No active enrollment of patients onto other PROS trials (practice)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rates of clinician delivering cessation assistance other than advice as assessed by parent surveys at baseline and 12 months after clinic visit
Rates of 7-day abstinence as confirmed biochemically at 12 months after clinic visit

SECONDARY OUTCOMES:
Rates of clinician asking about parental smoking as assessed by parent surveys at baseline and 12 months after clinic visit
Rates of clinician advising parents to quit as assessed by parent surveys at baseline and 12 months after clinic visit
Rates of clinician counseling parents about institution of rules prohibiting smoking in the home and car as assessed by parent surveys at baseline and 12 months after clinic visit
Percentage of parental smokers who have 7-day abstinence at both 3 and 12 months after clinic visit
Percentage of parental smokers reported quit attempts lasting at least 24 hours as assessed by parent surveys at baseline, 3 months, and 12 months after clinic visit
Percentage of parental smokers using pharmacotherapy (i.e., gum, patch, lozenge, inhaler, nasal spray, or bupropion) for smoking cessation as assessed by parent surveys at baseline, 3 months, and 12 months after clinic visit
Percentage of parental smokers who received telephone counseling or other services as assessed by parent surveys at baseline, 3 months, and 12 months after clinic visit
Percentage of parental smokers who instituted home and car smoking bans, as assessed by parent surveys at baseline, 3 months, and 12 months after clinic visit
Percentage of parental smokers who expose children to second-hand smoke as assessed by parent surveys at baseline, 3 months, and 12 months after clinic visit
Practice implementation of tobacco control office system as assessed by process survey of clinicians and key office staff at baseline and then at 6 weeks and 6 months after completion of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Winickoff, MD, MPH, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Drehmer JE, Hipple B, Ossip DJ, Nabi-Burza E, Winickoff JP. A Cross-Sectional Study of Happiness and Smoking Cessation among Parents. J Smok Cessat. 2017 Mar;12(1):6-14. doi: 10.1017/jsc.2015.6. Epub 2015 Mar 24. PMID 28163788
- [Derived] Drehmer JE, Hipple B, Nabi-Burza E, Ossip DJ, Chang Y, Rigotti NA, Winickoff JP. Proactive enrollment of parents to tobacco quitlines in pediatric practices is associated with greater quitline use: a cross-sectional study. BMC Public Health. 2016 Jun 24;16:520. doi: 10.1186/s12889-016-3147-1. PMID 27342141
- [Derived] Winickoff JP, Nabi-Burza E, Chang Y, Regan S, Drehmer J, Finch S, Wasserman R, Ossip D, Hipple B, Woo H, Klein J, Rigotti NA. Sustainability of a parental tobacco control intervention in pediatric practice. Pediatrics. 2014 Nov;134(5):933-41. doi: 10.1542/peds.2014-0639. Epub 2014 Oct 20. PMID 25332492
- [Derived] Mahabee-Gittens EM, Collins BN, Murphy S, Woo H, Chang Y, Dempsey J, Weiley V, Winickoff JP. The parent-child dyad and risk perceptions among parents who quit smoking. Am J Prev Med. 2014 Nov;47(5):596-603. doi: 10.1016/j.amepre.2014.07.010. Epub 2014 Sep 4. PMID 25201508
- [Derived] Drehmer JE, Ossip DJ, Nabi-Burza E, Rigotti NA, Hipple B, Woo H, Chang Y, Winickoff JP. Thirdhand smoke beliefs of parents. Pediatrics. 2014 Apr;133(4):e850-6. doi: 10.1542/peds.2013-3392. Epub 2014 Mar 3. PMID 24590745
- [Derived] Winickoff JP, Nabi-Burza E, Chang Y, Finch S, Regan S, Wasserman R, Ossip D, Woo H, Klein J, Dempsey J, Drehmer J, Hipple B, Weiley V, Murphy S, Rigotti NA. Implementation of a parental tobacco control intervention in pediatric practice. Pediatrics. 2013 Jul;132(1):109-17. doi: 10.1542/peds.2012-3901. PMID 23796741
- [Derived] Friebely J, Rigotti NA, Chang Y, Hall N, Weiley V, Dempsey J, Hipple B, Nabi-Burza E, Murphy S, Woo H, Winickoff JP. Parent smoker role conflict and planning to quit smoking: a cross-sectional study. BMC Public Health. 2013 Feb 22;13:164. doi: 10.1186/1471-2458-13-164. PMID 23433098
- [Derived] Drehmer JE, Ossip DJ, Rigotti NA, Nabi-Burza E, Woo H, Wasserman RC, Chang Y, Winickoff JP. Pediatrician interventions and thirdhand smoke beliefs of parents. Am J Prev Med. 2012 Nov;43(5):533-6. doi: 10.1016/j.amepre.2012.07.020. PMID 23079177